CLINICAL TRIAL: NCT01190397
Title: Phase I, Prospective, Comparative Study, Investigator Masked , Monocentric Measuring Warming Efficiency and Safety of Blephasteam® Versus Warm Compresses in Eyelid Therapy
Brief Title: Warming Efficiency of Warm Compresses Versus BLEPHASTEAM® in Eyelid Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LT2420-PI-CE-07/10
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Eyelid Diseases
Keywords: Warming goggles
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blephasteam Arm (Experimental)
  Interventions: Device: Warming goggles
- warm and moist compresses arm (Active Comparator)
  Interventions: Device: warm and moist compresses

INTERVENTIONS:
Device: Warming goggles
  Arms: Blephasteam Arm
Device: warm and moist compresses
  Arms: warm and moist compresses arm

SUMMARY:
The eyelid warming device is designed to relieve the symptoms of dysfunction of the glands in the eyelids

Phase I, prospective, comparative study, investigator masked , monocentric

Objectives are To assess and compare the warming and moisture of Blephasteam® device versus the warming and moisture of warm and moist compresses.

To assess and compare safety on the ocular surface after 10 minutes of Blephasteam® application versus after 10 minutes of warm and moist compresses application

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 80 years old.
* Healthy volunteers.
* For any contact lens wearers, they must be wearing hydrogel contact lenses (worn at least 3 times per week)
* Normal ocular examination in both eyes.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Temperature measurements
  The temperature in the chamber of the goggles for Blephasteam device, or between the lid and the compresses for the moist and warm compress, will be evaluated in 10 consecutive measurements over a period of 10 minutes with a micro sensor at the lower lid margin of one randomly selected eye of 10 randomly selected subjects

SECONDARY OUTCOMES:
Humidity measurements
  The humidity in the chamber of the goggles for Blephasteam device, or between the lid and the compresses for the moist and warm compress, will be evaluated in 10 consecutive measurements over a period of 10 minutes with a micro sensor at the lower lid margin of one randomly selected eye of 10 randomly selected subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Heiko PULT, Doctor, Principal Investigator — Cardiff University
Locations (1):
- School of Optometry & Vision Sciences, Cardiff, United Kingdom